CLINICAL TRIAL: NCT01630616
Title: A Single-Dose Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Odanacatib in Adolescents and Young Adults Treated With Glucocorticoids
Brief Title: A Study of Odanacatib When Administered to Adolescents and Young Adults Treated With Glucocorticoids (MK-0822-066)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0822-066; MK-0822-066 (Other: Protocol Number)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Adolescents Odanacatib 10 mg (Experimental): Study drug (single oral dose of odanacatib 10 mg) was administered following at least an 8-hour fast to adolescents.
  Interventions: Drug: Odanacatib
- Adolescents Odanacatib 50 mg (Experimental): Study drug (single oral dose of odanacatib 50 mg) was administered following at least an 8-hour fast to adolescents.
  Interventions: Drug: Odanacatib
- Adolescents Placebo (Placebo Comparator): Study drug (single oral dose of placebo) was administered following at least an 8-hour fast to adolescents.
  Interventions: Drug: Placebo
- Young Adults Odanacatib 50 mg (Experimental): Study drug (single oral dose of odanacatib 50 mg) was administered following at least an 8-hour fast to young adults.
  Interventions: Drug: Odanacatib
- Young Adults Placebo (Placebo Comparator): Study drug (single oral dose of placebo) was administered following at least an 8-hour fast to young adults.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Odanacatib — single oral dose, tablets, 10 or 50 mg
  Other Names: MK-0822
  Arms: Adolescents Odanacatib 10 mg; Adolescents Odanacatib 50 mg; Young Adults Odanacatib 50 mg
Drug: Placebo — single oral dose, tablets
  Arms: Adolescents Placebo; Young Adults Placebo

SUMMARY:
This study will assess the safety, tolerability, pharmacodynamics, and pharmacokinetics of single doses of odanacatib in mature adolescents and young adults who are currently receiving glucocorticoid therapy. The primary hypotheses for the study are that a single dose of odanacatib is well tolerated in mature adolescents and following single dose administration of odanacatib 50 mg, there is no clinically important difference in AUC0-inf between mature adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of reproductive potential (or other female subjects at the discretion of the investigator) must have negative serum pregnancy test and agree to use (and/or have their partner use) two (2) acceptable methods of birth control beginning at the prestudy visit throughout the study and until 2 weeks after the dose of study
* Receiving glucocorticoid therapy at a dose anticipated to be stable over the course of the study period
* X-ray evidence of closed epiphyses (growth plate) at the hand
* Nonsmoker

Exclusion Criteria:

* Pregnant or unwilling to undergo pregnancy test
* History of stroke, chronic seizures, or major neurological disorder
* History of malignant neoplastic disease (cancer)
* Breastfeeding
* Primary growth disorder
* Any disease affecting the stomach or proximal small intestine resulting in malabsorption
* Received treatment which might have influenced bone turnover, including anabolic steroids, testosterone, calcitonin, calcitriol, alfacalcidol, excess vitamin A or excess vitamin D, or cyclosporine or initiation of use of birth control pills (estrogen-progestin combinations or progestin only, or depo provera) or other estrogen containing medications, or thyroid hormone unless on a stable dose for at least 1 month and has a normally functioning thyroid gland
* Previous treatment with any marketed or experimental bisphosphonate within 12 months
* History of, or evidence for, any clinically relevant metabolic bone disease (other than glucocorticoid-induced bone loss) including but not limited to primary hyperparathyroidism, hypoparathyroidism, hyperthyroidism, osteomalacia, and osteogenesis imperfecta within previous 3 years
* History of hypothyroidism
* Consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL), or participated in another investigational study within 4 weeks
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Regular user (including "recreational use") of any illicit drugs, or has a history of drug or alcohol abuse
* Unable to swallow tablets

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2016-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment continued until the Odanacatib Development Program was discontinued on 02-Sep-2016. No participants were actively receiving treatment at the time of study discontinuation.
Pre-assignment Details: The Young Adults Odanacatib 10 mg arm represents historical data from a separate study (MK-0822-007). As such, these participants were not enrolled in any part of the current MK-0822-066 study.
Groups:
- Young Adults Odanacatib 10 mg: Study drug (single oral dose of odanacatib 10 mg) was administered following at least an 8-hour fast to young adults (historical study MK-0822-007).
Period: Overall Study
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo
Started | 5 | 3 | 3 | 12 | 6 | 2
Completed | 5 | 3 | 3 | 9 | 6 | 2
Not Completed | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis of baseline characteristics are the participants used for the pharmacokinetic and statistical analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo | Total
Number analyzed (Participants) | 5 | 3 | 3 | 9 | 6 | 2 | 28
Age, Continuous [Mean (Full Range); unit: Years] | 14.8 (1.6) [13 to 16] | 15.7 (0.6) [15 to 16] | 16.3 (0.6) [16 to 17] | 26.6 (1.6) [19 to 37] | 22.3 (0.0) [20 to 24] | 20 [20 to 20] | 20.8 (3.4) [13 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 1 | 3 | 2 | 13
  Male | 1 | 1 | 2 | 8 | 3 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Report an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Day 14
Population: The population analyzed consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 3 | 3 | 6 | 2
Participants | 1 | 0 | 0 | 1 | 0

2. Primary Outcome: Area Under the Plasma-Drug Concentration Time Curve From Hour 0 to Infinity (AUC0-inf) For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 50 mg
Description: Area Under the Plasma-Drug Concentration/Time Curve from Time 0 to infinity (AUC0-inf) is a measure of the total amount of drug in the plasma from the dose administration to the last measurable sample. The Method of Dispersion is more accurately described as "Percent Geometric Coefficient of Variation". Pharmacokinetic (PK) analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 50 mg, who had available AUC0-inf data from at least one treatment. PK parameters were not analyzed for the Placebo arms and data are presented for the Adolescents Odanacatib 10 mg arm in other outcome measures.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 6 | 0
μM·hr |  | 21.6 (30.7) |  | 27.2 (40.4) |

3. Primary Outcome: Area Under the Plasma-Drug Concentration Time Curve From Hour 0 to 168 Hours (AUC0-168) For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 50 mg
Description: Area Under the Plasma-Drug Concentration/Time Curve from Time 0 to Hour 168 (AUC0-168) is a measure of the total amount of drug in the plasma from the dose administration to the Hour 168 sample. The Method of Dispersion is more accurately described as "Percent Geometric Coefficient of Variation". PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, and 168 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 50 mg, who had available AUC0-168 data from at least one treatment. PK parameters were not analyzed for the Placebo arms and data are presented for the Adolescents Odanacatib 10 mg arm in other outcome measures.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 6 | 0
μM·hr |  | 18.7 (24.0) |  | 21.5 (39.8) |

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Odanacatib For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 50 mg
Description: Cmax is a measure of the maximum amount of drug in the plasma after the drug dose is given. The Method of Dispersion is more accurately described as "Percent Geometric Coefficient of Variation". PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 50 mg, who had available Cmax data from at least one treatment. PK parameters were not analyzed for the Placebo arms and data are presented for the Adolescents Odanacatib 10 mg arm in other outcome measures.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 6 | 0
nM |  | 256 (30.8) |  | 237 (51.1) |

5. Primary Outcome: Time to Cmax (Tmax) of Odanacatib For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 50 mg
Description: Tmax is the time required to reach Cmax. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 50 mg, who had available Tmax data from at least one treatment. PK parameters were not analyzed for the Placebo arms and data are presented for the Adolescents Odanacatib 10 mg arm in other outcome measures.
Measure: Median (Full Range); unit: Hours
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 6 | 0
Hours |  | 6.0 [2.0 to 24.0] |  | 9.0 [1.0 to 24.0] |

6. Primary Outcome: Apparent Terminal Half-life (t1/2) of Odanacatib For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 50 mg
Description: T1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 50 mg, who had available t1/2 data from at least one treatment. PK parameters were not analyzed for the Placebo arms and data are presented for the Adolescents Odanacatib 10 mg arm in other outcome measures.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 6 | 0
Hours |  | 66.9 (30.4) |  | 77.3 (20.9) |

7. Secondary Outcome: Change From Baseline in Urinary Aminoterminal Crosslinked Telopeptide of Type 1 Collagen (uNTx/Cr) at 168 Hours Postdose
Description: Urinary aminoterminal crosslinked telopeptide of Type I collagen (uNTx/Cr) is a biochemical marker of bone resorption. Odanacatib selectively and potently inhibits cathepsin K (CatK), the primary catalyst of bone resorption. Since CatK is the enzyme responsible for bone matrix degradation it is possible to use bone resorption biomarkers to quantify pharmacodynamic effects in short term clinical studies. CatK cleaves the N-telopeptide of collagen type I to form NTx and also cleaves the serum C-terminal telopeptide of collagen type I (1-CTP - itself generated by the action of matrix metalloproteases) to generate CTx. Urine NTx measurements (in bone collagen equivalents [BCE]) have been normalized to creatinine clearance.
Time Frame: Baseline (predose Day 1) and 168 hours postdose
Population: The population analyzed included all randomized, treated participants who had available uNTx/Cr data for Baseline and 168 hours.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol[BCE]/mmol[creatinine])
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 3 | 3 | 6 | 2
nmol[BCE]/mmol[creatinine]) | 0.79 (50.68) | 0.40 (232.0) | 1.03 (3.39) | 0.36 (53.62) | 0.83 (13.53)

8. Primary Outcome: AUC0-inf for Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 10 mg
Description: Area Under the Plasma Concentration/Time Curve from Time 0 to infinity (AUC0-inf) is a measure of the total amount of drug in the plasma from the dose administration to the last measurable sample. The AUC0-inf data for 10 mg odanacatib in adolescents were compared with the historical young adult odanacatib 10 mg AUC0-inf data from study MK-0822-007. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 10 mg, who had available AUC0-inf data from at least one treatment including young adults from historical study MK-0822-007. PK parameters were not analyzed for the Placebo arms and data are presented for the Odanacatib 50 mg arms in other outcome measures.
Measure: Geometric Mean (95% Confidence Interval); unit: μM·hr
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 0 | 0 | 9 | 0 | 0
μM·hr | 10 [7.5 to 13.3] |  |  | 11.3 [9.1 to 13.9] |  |
Statistical Analysis 1: Comparison: Adolescents Odanacatib 10 mg vs Young Adults Odanacatib 10 mg; Test type: Superiority or Other; Ratio (Adolescents/adults) = 0.89, 90% CI 2-sided [0.62 to 1.26]

9. Primary Outcome: AUC0-168 for Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 10 mg
Description: Area Under the Plasma Concentration/Time Curve from Time 0 to Hour 168 (AUC0-168) is a measure of the total amount of drug in the plasma from the dose administration to the Hour 168 sample. The AUC0-168 data for 10 mg odanacatib in adolescents were compared with the historical young adult odanacatib 10 mg AUC0-168 data from study MK-0822-007. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, and 168 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 10 mg, who had available AUC0-168 data from at least one treatment including young adults from historical study MK-0822-007. PK parameters were not analyzed for the Placebo arms and data are presented for the Odanacatib 50 mg arms in other outcome measures.
Measure: Geometric Mean (95% Confidence Interval); unit: μM·hr
Groups:
- Adolescents Odanacatib 50: Study drug (single oral dose of odanacatib 50 mg) was administered following at least an 8-hour fast to adolescents.
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 0 | 0 | 9 | 0 | 0
μM·hr | 8.1 [6.2 to 10.7] |  |  | 9.3 [7.6 to 11.4] |  |
Statistical Analysis 1: Comparison: Adolescents Odanacatib 10 mg vs Young Adults Odanacatib 10 mg; Test type: Superiority or Other; Ratio (Adolescents/Adults) = 0.87, 90% CI 2-sided [0.62 to 1.23]

10. Primary Outcome: Cmax of Odanacatib For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 10 mg
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. The Cmax data for 10 mg odanacatib in adolescents were compared with the historical young adult odanacatib 10 mg Cmax data from study MK-0822-007. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 10 mg, who had available Cmax data from at least one treatment including young adults from historical study MK-0822-007. PK parameters were not analyzed for the Placebo arms and data are presented for the Odanacatib 50 mg arms in other outcome measures.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 0 | 0 | 9 | 0 | 0
nM | 99.6 [75.0 to 132.4] |  |  | 122.3 [99.0 to 151.1] |  |
Statistical Analysis 1: Comparison: Adolescents Odanacatib 10 mg vs Young Adults Odanacatib 10 mg; Test type: Superiority or Other; Ratio (Adolescents/Adults) = 0.81, 90% CI 2-sided [0.57 to 1.16]

11. Primary Outcome: Tmax of Odanacatib For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 10 mg
Description: Tmax is the time required to reach Cmax. The Tmax data for 10 mg odanacatib in adolescents were compared with the historical young adult odanacatib 10 mg Tmax data from study MK-0822-007. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 10 mg, who had available Tmax data from at least one treatment including young adults from historical study MK-0822-007. PK parameters were not analyzed for the Placebo arms and data are presented for the Odanacatib 50 mg arms in other outcome measures.
Measure: Median (Full Range); unit: Hours
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 0 | 0 | 9 | 0 | 0
Hours | 6.0 [6.0 to 24.0] |  |  | 6.0 [4.0 to 32.0] |  |

12. Primary Outcome: Apparent Terminal t1/2 of Odanacatib For Adolescents and Young Adults Following a Single Oral Dose of Odanacatib 10 mg
Description: Apparent terminal t1/2 is the time required for a given drug concentration in the plasma to decrease by 50%. The apparent terminal t1/2 data for 10 mg odanacatib in adolescents were compared with the historical young adult odanacatib 10 mg apparent terminal t1/2 data from study MK-0822-007. PK analysis was not performed on participants receiving placebo.
Time Frame: Hour 0 (predose), and at 1, 2, 6, 8, 12, 24, 72, 96, 120, 168, 240, and 336 hours post-dose
Population: The population analyzed included all randomized participants, treated with odanacatib 10 mg, who had available t1/2 data from at least one treatment including young adults from historical study MK-0822-007. PK parameters were not analyzed for the Placebo arms and data are presented for the Odanacatib 50 mg arms in other outcome measures.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 10 mg | Young Adults Odanacatib 50 mg | Young Adults Placebo
Number analyzed (Participants) | 5 | 0 | 0 | 9 | 0 | 0
Hours | 80.5 (17.9) |  |  | 73.0 (23.4) |  |

ADVERSE EVENTS:
Time Frame: Up to Day 14 (MK-0822-066) & Up to 408 hours post-dose (historical study MK-0822-007)
Description: The population analyzed consisted of all randomized participants who received at least 1 dose of study drug. The Young Adults Odanacatib 10 mg arm represent historical data from a separate study (MK-0822-007). As such, these participants were not enrolled in any part of the current MK-0822-066 study.
Arm/Group | Adolescents Odanacatib 10 mg | Adolescents Odanacatib 50 mg | Adolescents Placebo | Young Adults Odanacatib 50 mg | Young Adults Placebo | Young Adults Odanacatib 10 mg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/3 | 0/6 | 0/2 | 0/12
Other Adverse Events (participants affected / at risk) | 1/5 | 0/3 | 0/3 | 1/6 | 0/2 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents Odanacatib 10 mg (N=5) | Adolescents Odanacatib 50 mg (N=3) | Adolescents Placebo (N=3) | Young Adults Odanacatib 50 mg (N=6) | Young Adults Placebo (N=2) | Young Adults Odanacatib 10 mg (N=12)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.